CLINICAL TRIAL: NCT03332550
Title: A National, Registry Based Study of Clinical Results After Emergency Operation for Perforated Diverticulitis to Compare Laparoscopic Lavage and Resection Surgery in Routine Use.
Brief Title: A National Study of Clinical Results After Emergency Operation for Perforated Diverticulitis
Acronym: LapLav
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Haglind, MD, PhD, professor, MD, PhD, professor, Sahlgrenska University Hospital
Other Study IDs: LapLav
Record Dates: First submitted 2017-10-10; First posted 2017-11-06 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Perforated Diverticulitis
Keywords: laparoscopic lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- purulent peritonitis: Hinchey 3
  Interventions: Procedure: Laparoscopic lavage; Procedure: Colon resection
- faecal peritonitis: Hinchey 4
  Interventions: Procedure: Colon resection

INTERVENTIONS:
Procedure: Laparoscopic lavage — Operation with laparoscopic lavage for perforated diverticulitis Hinchey 3
  Groups: purulent peritonitis
Procedure: Colon resection — Operation with colon resection for perforated diverticulitis Hinchey 4

SUMMARY:
The aim of this study is to evaluate clinical results and effect on health and well-being in patients operated for perforated diverticulitis with purulent peritonitis by laparoscopic lavage in Sweden when used outside of prospective studies/trials and in comparison with the traditional treatment, i.e. colon resection with or without stoma formation.

A secondary aim is to evaluate the outcome after fecal peritonitis.

The hypothesis is that laparoscopic lavage as treatment for perforated diverticulitis with purulent peritonitis is safe, efficient and cost saving, when used in routine health care.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered in the Patient registry with ICD 10 codes K57 classified as emergency admissions and with the Nordic Medico-Statistical Committee (NOMESCO) code JAH01(diagnostic laparoscopy), JFB46 (resection of sigmoid colon), JFB60 (resection of sigmoid colon, sigmoidostomy and closure of the distal stump), JFB61 (laparoscopic resection of sigmoid colon, sigmoidostomy and closure of the distal stump), JFB63 (other colon resection, colostomy and closure of the distal stump), JAK04 (laparoscopy and peritoneal lavage), JAW97 (other laparoscopic operation involving abdominal wall, mesentery, peritoneum or the omentum)

Exclusion Criteria:

* Patients where hospital records reveal that the index admission was misclassified (not perforated diverticulitis) will be excluded.
* Patients classified as Hinchey 1-2.
* No informed consent received or withdrawal of consent (questionnaire)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All swedish patients registrered within the Swedish Patient Registry with ICD 10 codes K57 classified as emergency admissions and with a NOMESCO code JAH01, JFB46 , JFB60, JFB61, JFB63, JAK04, JAW97.
  The cohort will be divided into two groups when analysing and presenting results, perforated diverticulitis with purulent peritonitis (Hinchey grade III) and perforated diverticulitis with faecal peritonitis (Hinchey grade IV) .
Sampling Method: Non-Probability Sample
Enrollment: 669 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Need for further surgical interventions within 12 months of index surgery | 12 months
  Number of patients in need of further surgical interventions within 12 months after index surgery.

SECONDARY OUTCOMES:
Need for further surgical interventions within 24 months of index surgery | 24 months
  Number of patients in need of further surgical interventions within 24 months after index surgery.
Colon cancer diagnosis | 12 months
  Number of colon cancer diagnosis within 12 months
Health economics with regard to the two different treatment modalities. | 2 years
  In the analysis data from the study will be combined with prices from the cost-per-patient system at Sveriges Kommuner och Landsting, or where appropriate, from Sahlgrenska University Hospital, in combination with sensitivity testing of results.
Percentages of all cases treated by laparoscopic lavage and emergency colon resection, respectively. | 36 months
  Percentages of all cases treated by laparoscopic lavage and emergency colon resection, respectively in a national Swedish cohort and in routine health care.
Complications (Clavien-Dindo ≥ IIIa) within 90 days of index surgery. | 90 days
  Complications (Clavien-Dindo ≥ IIIa) within 90 days of index surgery.
Mortality (90 days and 12 months respectively). | 12 months
  Mortality (90 days and 12 months respectively).
Patient reported outcome after treatment for perforated diverticulitis, function | 3 years
  Patient reported outcome as measured using a disease specific questionnaire 2-3 years after index surgery. The questionnaire is developed specifically for this study and will address prevalence, severity and associated distress of symptoms using Likert-type scales regarding function after surgery for perforated diverticulitis.
Patient reported outcome after treatment for perforated diverticulitis, quality of life | 3 years
  Patient reported outcome using a questionnaire sent out 2-3 years after index surgery for perforated diverticulitis, using EQ-5D for quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Haglind, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västa Götaland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angenete E, Bock D, Rosenberg J, Haglind E. Laparoscopic lavage is superior to colon resection for perforated purulent diverticulitis-a meta-analysis. Int J Colorectal Dis. 2017 Feb;32(2):163-169. doi: 10.1007/s00384-016-2636-0. Epub 2016 Aug 27. PMID 27567926
- [Background] Angenete E, Thornell A, Burcharth J, Pommergaard HC, Skullman S, Bisgaard T, Jess P, Lackberg Z, Matthiessen P, Heath J, Rosenberg J, Haglind E. Laparoscopic Lavage Is Feasible and Safe for the Treatment of Perforated Diverticulitis With Purulent Peritonitis: The First Results From the Randomized Controlled Trial DILALA. Ann Surg. 2016 Jan;263(1):117-22. doi: 10.1097/SLA.0000000000001061. PMID 25489672
- [Background] Gehrman J, Angenete E, Bjorholt I, Bock D, Rosenberg J, Haglind E. Health economic analysis of laparoscopic lavage versus Hartmann's procedure for diverticulitis in the randomized DILALA trial. Br J Surg. 2016 Oct;103(11):1539-47. doi: 10.1002/bjs.10230. Epub 2016 Aug 22. PMID 27548306
- [Background] Schultz JK, Wallon C, Blecic L, Forsmo HM, Folkesson J, Buchwald P, Korner H, Dahl FA, Oresland T, Yaqub S; SCANDIV Study Group. One-year results of the SCANDIV randomized clinical trial of laparoscopic lavage versus primary resection for acute perforated diverticulitis. Br J Surg. 2017 Sep;104(10):1382-1392. doi: 10.1002/bjs.10567. Epub 2017 Jun 20. PMID 28631827
- [Background] Vennix S, Musters GD, Mulder IM, Swank HA, Consten EC, Belgers EH, van Geloven AA, Gerhards MF, Govaert MJ, van Grevenstein WM, Hoofwijk AG, Kruyt PM, Nienhuijs SW, Boermeester MA, Vermeulen J, van Dieren S, Lange JF, Bemelman WA; Ladies trial colloborators. Laparoscopic peritoneal lavage or sigmoidectomy for perforated diverticulitis with purulent peritonitis: a multicentre, parallel-group, randomised, open-label trial. Lancet. 2015 Sep 26;386(10000):1269-1277. doi: 10.1016/S0140-6736(15)61168-0. Epub 2015 Jul 22. PMID 26209030
- [Background] Thornell A, Angenete E, Bisgaard T, Bock D, Burcharth J, Heath J, Pommergaard HC, Rosenberg J, Stilling N, Skullman S, Haglind E. Laparoscopic Lavage for Perforated Diverticulitis With Purulent Peritonitis: A Randomized Trial. Ann Intern Med. 2016 Feb 2;164(3):137-45. doi: 10.7326/M15-1210. Epub 2016 Jan 19. PMID 26784672
- [Derived] Samuelsson A, Bock D, Prytz M, Block M, Ehrencrona C, Wedin A, Angenete E, Haglind E. Functional Outcomes of Emergency Surgery for Perforated Diverticulitis, Hinchey Grade III. World J Surg. 2023 Jun;47(6):1570-1582. doi: 10.1007/s00268-023-06961-2. Epub 2023 Mar 1. PMID 36856835